CLINICAL TRIAL: NCT03088436
Title: Feasibility Study of Supine Breast MRI : Comparison With Prone MRI and Comfort Assessment
Status: Completed | Type: Observational
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Other Study IDs: ICL_2014_0003
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Breast Diseases
Keywords: MRI; Breast
MeSH Terms: conditions — Breast Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: preoperative prone MRI and supine second-look ultrasound data — Patients were examined using a standard clinical MRI protocol in the prone position with both arms placed above the head. Second-look ultrasonographies were performed. Patients were instructed to lie supine, with their hands behind their heads.

SUMMARY:
The aim of the present study was to determine the prone-to-supine displacement of breast lesions using preoperative prone MRI and supine second-look ultrasound data

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were being a woman with breast lesions whose assessment involved breast MRI and ultrasound at our institution. There were no exclusion criteria.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients records were extracted from the electronic health record system of Institut de Cancérologie de Lorraine
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

PRIMARY OUTCOMES:
distance to the nipple (mm) | 1 day
  the distance to the nipple for lesion was determined using prone MRI and supine ultrasound